CLINICAL TRIAL: NCT03349216
Title: Comparison of Intravenous Regional Anesthesia ( Bier's Block) and Systemic Analgesia for Upper Extremity Procedures in the Emergency Department of Al-Zahra University Hospital
Brief Title: Bier's Block Versus Systemic Analgesia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mehdi Nasr Isfahani, Clinical Professor, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 395608
Record Dates: First submitted 2017-11-11; First posted 2017-11-21 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures | interventions — Conscious Sedation

STUDY DESIGN:
Intervention Model Description: Bier's Block with Lidocaine versus Conscous Sedation with ketamine
Masking Description: not blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous regional Analgesia (Experimental): in this arm patients will receive intravenous regional anesthesia as infusion of mini dose (that is 1.5 mg/kg ) lidocaine 0.5% and immediately after procedure their torniquettes will be deflated (hence named Rapid MiniBier's block).
  Interventions: Procedure: Intravenous Regional Anesthesia
- Systemic Analgesia (Experimental): In this arm patients will receive ketamine 1-2 mg/kg IV slow as a systemic analgesia. ketamine as a PCP derivative has both hypnotic and analgesic effects.
  Interventions: Drug: Systemic Analgesia

INTERVENTIONS:
Procedure: Intravenous Regional Anesthesia — in this research patients will receive intravenous regional anesthesia as infusion of mini dose (that is 1.5 mg/kg ) lidocaine 0.5% and immediately after procedure their torniquettes (A.T.S. 2000, Zimmer, Inc., Bloomfield, CN) will be deflated (hence named Rapid MiniBier's block). the pain score will be assessed by NRS system before during and after the procedure.
  Other Names: Bier's Block
  Arms: Intravenous regional Analgesia
Drug: Systemic Analgesia — in this group the patients will receive ketamine 1-2 mg/kg IV slow ( Bioniche,Ireland Ketamine Hydrochloride 500mg/10cc)and titrated to effect. again here the pain score will be assessed before procedure and after the procedure every 5 minutes until 30 minutes by NRS ( Numerical Rating Score)
  Other Names: Conscious Sedation
  Arms: Systemic Analgesia

SUMMARY:
Background: There are three methods for procedural sedation in upper extremity traumas; systemic, regional and local anesthesia. There is controversy in the literature regarding the method of choice for this purpose.

Objectives: The aim of this study was to compare conscious sedation and Bier's block methods for pain reduction in upper extremity trauma patients.

Patients and Methods: This was a randomized clinical trial. Patients were randomly allocated to either the Bier's block or the conscious sedation group. Pain reduction was assessed by a numerical rating scale; patients, surgeons and physicians responsible for analgesia satisfaction were assessed using a five-point Likert scale.

In this study, we aimed to compare the effectiveness, complications, duration, hemodynamic stability and patient and physician satisfaction between systemic analgesia and Bier's block method performed at the emergency department.

DETAILED DESCRIPTION:
Patients and Methods

Study Design

This is a randomized clinical trial to be conducted at two tertiary health care centers, with census of 102000 and 60000 visits per year, during years 2017 and 2018. The study design has been approved by ethics committee of the university. Informed consents will be obtained from patients. And patients who refuse to participate in the study are excluded from the study and will receive analgesia based on the physician responsible for analgesia preference.

Population

All adult patients (aged 18 or more) with upper extremity trauma who need procedural analgesia in the ED are included in this study. Patients with a history of seizure, known allergy to analgesic substances, sickle cell anemia, peripheral vascular disease and arteriovenous fistula or infection in upper extremities are excluded from the study. Patients who need emergent intervention/s that last more than one hour are also excluded from the study. Randomization is done using sealed envelopes containing computer-generated block random allocation numbers.

Intervention

After introduction of the protocol of Bier's block (using 1.5 mg/kg of 0.5% lidocaine) or systemic analgesia (using ketamine 1.5 mg/kg), patients underwent the necessary procedure. Physicians who were responsible for the analgesia, had authority to change the method of analgesia in each group, if necessary.

Measurements

Patient's age, sex, site and type of injury, vital signs and pain score using the Numerical Rating Scale (NRS) will be recorded before the introduction of analgesia. Patient's vital signs are documented at the end of the procedure. Satisfaction of the patient, surgeon and physician responsible for analgesia for the applied analgesic method is obtained before discharge from the ED operating room. Patients also score their level of pain before discharge and their vital signs are recorded at another instance. Time of initiation of analgesia, initiation of procedure, end of procedure, and gaining consciousness in systemic analgesia group and time of discharge from ED operating room are documented and patients will be discharged from the ED operating room when eligible.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (aged 18 or more) with upper extremity trauma who need procedural analgesia

Exclusion Criteria:

* Patients with a history of seizure
* Known allergy to analgesic substances
* Sickle cell anemia,
* Peripheral vascular disease and arteriovenous fistula
* Infection in upper extremities
* Patients who need emergent intervention/s that last more than one hour are also excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
pain score | 30 minutes since the beginning of procedure
  pain score assessed as numerical analogue score (NRS) with 1 for minimum and 10 for the maximum pain experienced by patient. A decrease of at least 13 millimeter will be considered as statistically meaningful.

SECONDARY OUTCOMES:
Complications | 30 minutes
  Seizure

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Nasr Isfahani, M.D., Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Al-Zahra Hospital, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Isfahani MN, Naseh K, Golshani K. Mini-dose Bier's block vs systemic analgesia in distal radius fractures: a promising reduction in emergency department throughput time. Pain Manag. 2023 Aug;13(8):433-443. doi: 10.2217/pmt-2023-0030. Epub 2023 Sep 18. PMID 37718930